CLINICAL TRIAL: NCT04349904
Title: Near-Focus Narrow Band Imaging Classification of Villous Atrophy in Suspected Coeliac Disease: International Development and Validation
Brief Title: Near-Focus NBI Classification of Villous Atrophy in Suspected Coeliac Disease: International Development and Validation
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Olympus (Industry)
Responsible Party: Sponsor
Other Study IDs: 222807
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — duodenal samples for histopathological evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Near-Focus Narrow Band Imaging — High Definition White Light Endoscopic Imaging followed by Near-Focus Narrow Band Imaging and target biopsy of 6 areas of the duodenum (2 from the first part and 4 from the second part of the duodenum)

SUMMARY:
There are no agreed endoscopic signs for the diagnosis of villous atrophy(VA) in coeliac disease(CD), necessitating biopsies and for both diagnosis and exclusion. Here we evaluated the role of near focus Narrow Band Imaging(NF-NBI) for the assessment of villous architecture in suspected CD with development and further validation of a novel NF-NBI classification.

DETAILED DESCRIPTION:
Coeliac disease (CD) is an autoimmune condition by the exposure to gluten in patients who are genetically susceptible. The global prevalence is thought to be 1%, and incidence rate of CD in the UK is approximately 13.8 per 100,000 person-years with greater than fourfold increase in incidence over the past two decades [1]. CD has variable clinical presentations including iron deficiency anaemia, diarrhoea, bloating, weight loss, osteoporosis, rash and rarely lymphoma. The ingestion of gluten triggers an immune response with the production of antibodies and an inflammatory destruction of small bowel (duodenal) mucosa (villous atrophy). The degree of villous atrophy is categorised based on duodenal biopsy analysis according to the Marsh classification [2]. Serological testing for antibody formation has varying sensitivity and specificity for CD with extent of villous damage [3]. At present the diagnosis of CD required confirmation on histopathological analysis of duodenal biopsy [4]. The British Society of Gastroenterology (BSG) requires the investigation of CD in all patients with iron deficiency anaemia as well as other symptoms above suggestive of CD [5]. Gastroscopy and duodenal biopsies are the current gold standard for exclusion or confirmation of CD [6]. Examination with standard white light endoscopy (WLE) can reveal patchy redness (erythema) of the small bowel mucosa and possibly appearance of flattening of the duodenal villi however due to limited sensitivity especially in milder cases of villous distortion and atrophy, biopsy is warranted [7]. Owing to this patchy nature of villous atrophy, orientation of biopsy is also imperative for accurate diagnosis of CD including biopsies from the duodenal bulb as well as the second part of the duodenum [8,9]. Although biopsy is the gold standard for diagnosis of CD, it is limited by inadequate quality and orientation of sampling contributing to false negative [10]. Various endoscopic imaging techniques have been studied for the diagnosis of CD by assessment of villous architecture. The water immersion technique involves filling the lumen of the duodenum with water has shown promising sensitivity and specificity for the diagnosis of CD. Further study to assess reproducibility are warranted [11,12]. Magnification endoscopy has demonstrated reasonable positive and negative predictive value with a fair degree of reproducibility within the remit of preliminary data [13]. The addition of agents to enhance villous architecture during endoscopic examination such a water soluble blue dye spray (chromendoscopy) or ascetic acid have been assessed. Chromendoscopy has shown promising sensitivity and specificity for CD, however it has not been consistently demonstrated to be superior to WLE alone and no further benefit achieved when combining chromendoscopy to magnification endoscopy [14,15]. Furthermore, chromendoscopy is limited by operator technical ability in achieving a uniform coating of dye, interpretation and prolongs time and cost [16]. The addition of ascetic acid increased sensitivity for detecting villous atrophy and demonstrating the patchy nature of this to aid target biopsy but there is insufficient evidence to support the use of this for endoscopic diagnosis of CD alone [17]. Preliminary data for digital imaging technology; virtual chromendoscopy provided by Fujinon Intelligent Chromo Endoscopy (FICE) and i-scan developed by Pentax Medical, Japan have been conducted for the diagnoses of CD. FICE with magnification has shown 100% accuracy for evaluating villous patterns and i-scan for the diagnosis of total villous atrophy using I-scan but studies demonstrating reproduction of this have not been conducted [18,19]. Narrow Band Imaging (NBI) provides an IEE technique unique to Olympus Medical Systems. NBI provides unique images based on penetrative properties of light in tissue which is directly proportional to wavelength with a use of a filter integral to the endoscope which is switched on using a button on the hand control at the time of examination. This filter produces two narrow bands at specific wavelengths; 415nm blue light and 540nm green light which is absorbed by superficial and deep mucosal vessels respectively. NBI provides a distinct contrast between vascular architecture and mucosa as NBI wavelength is reflected by mucosa but absorbed by blood vessels and has been shown to add diagnostic value in a variety of diagnostic settings most notably in the distinction between neoplastic and non-neoplastic lesions of the gastrointestinal tract [20]. It is the distortion of the villous vascular pattern as seen with varying degrees of villous atrophy that has the potential of making an optical diagnosis of coeliac disease even in its early stages, obviating the need for routine biopsy [9]. Clear endoscopic images of villous atrophy in comparison to healthy villi have been published using high resolution narrow band imaging in known CD [21]. Preliminary study of magnification in combination with NBI has shown feasibility for the detection of both total villous and partial villous atrophy, superiority to WLE with observer agreement [22,23]. A prospective observational study assessing the use of narrow band imaging in assessing duodenal villous atrophy in a variety of clinical scenarios has been performed however patients with a known diagnosis of coeliac disease were excluded [24,25]. These studies are limited by small sample size with only preliminary data for inter-observer variation. Dual focus NBI is a unique imaging system to Olympus endoscopic technology involving two-stage optical system operated by a single push of a button on the controller. The 'near' mode provides higher resolution power compared to previous NBI generations and holds enhanced brightness and contrast ability. This study will assess the ability of dual focus NBI for the endoscopic diagnosis of coeliac disease. To date there are no large prospective observational cohort studies evaluating conventional endoscopy and dual focus narrow band imaging for the endoscopic diagnosis and assessment of coeliac disease. Additionally there is limited data on inter-observer variation using NBI across degrees of endoscopic expertise; an important consideration when translating research findings to wide clinical practice. Additionally, NBI is readily available in most UK endoscopy centres making its implementation in practice relatively straightforward and of limited financial implication.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-90 years old
* Retaining capacity and medically fit for gastroscopy
* Requiring gastroscopy by current BSG guidelines for the investigation of anaemia or symptoms to suggest CD or positive serology.
* Assessment of CD

Exclusion Criteria:

* Outside inclusion age range
* Unable to give informed consent
* Clinical indication not satisfying inclusion criteria

Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients attending the gastroenterology department requiring gastroscopy and duodenal biopsy to evaluate Villous Atrophy (VA) were approached for recruitment. All patients were recruited who satisfied British Society of Gastroenterology (BSG) criteria for the investigation of suspected Coeliac Disease (CD): positive coeliac serology, iron deficiency anaemia, weight loss, bloating, diarrhoea
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2019-02-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the diagnostic performance of Near-Focus NBI (NF-NBI) for the diagnosis and assessment of Villous Atrophy (VA) in suspected Coeliac Disease (CD). | 6 weeks post endoscopy and duodenal biopsy
  Sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value, Accuracy

SECONDARY OUTCOMES:
To develop and initially validate a novel NF-NBI classification of VA | 3 months post completion of data collection
  Sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value, Accuracy, Inter-observer agreement

CONTACTS AND LOCATIONS:
Overall Officials: Bu'Hussain Hayee, FRCP PhD, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Shared upon request

REFERENCES:
- [Background] West J, Fleming KM, Tata LJ, Card TR, Crooks CJ. Incidence and prevalence of celiac disease and dermatitis herpetiformis in the UK over two decades: population-based study. Am J Gastroenterol. 2014 May;109(5):757-68. doi: 10.1038/ajg.2014.55. Epub 2014 Mar 25. PMID 24667576
- [Background] Marsh MN. Gluten, major histocompatibility complex, and the small intestine. A molecular and immunobiologic approach to the spectrum of gluten sensitivity ('celiac sprue'). Gastroenterology. 1992 Jan;102(1):330-54. PMID 1727768
- [Background] Rostom A, Dube C, Cranney A, Saloojee N, Sy R, Garritty C, Sampson M, Zhang L, Yazdi F, Mamaladze V, Pan I, McNeil J, Moher D, Mack D, Patel D. Celiac disease. Evid Rep Technol Assess (Summ). 2004 Jun;(104):1-6. No abstract available. PMID 15346868
- [Background] Goddard AF, James MW, McIntyre AS, Scott BB; British Society of Gastroenterology. Guidelines for the management of iron deficiency anaemia. Gut. 2011 Oct;60(10):1309-16. doi: 10.1136/gut.2010.228874. Epub 2011 May 11. PMID 21561874
- [Background] Rubio-Tapia A, Hill ID, Kelly CP, Calderwood AH, Murray JA; American College of Gastroenterology. ACG clinical guidelines: diagnosis and management of celiac disease. Am J Gastroenterol. 2013 May;108(5):656-76; quiz 677. doi: 10.1038/ajg.2013.79. Epub 2013 Apr 23. PMID 23609613
- [Background] Dickey W. Endoscopic markers for celiac disease. Nat Clin Pract Gastroenterol Hepatol. 2006 Oct;3(10):546-51. doi: 10.1038/ncpgasthep0601. PMID 17008924
- [Background] Hopper AD, Cross SS, Sanders DS. Patchy villous atrophy in adult patients with suspected gluten-sensitive enteropathy: is a multiple duodenal biopsy strategy appropriate? Endoscopy. 2008 Mar;40(3):219-24. doi: 10.1055/s-2007-995361. Epub 2008 Dec 5. PMID 18058655
- [Background] Cammarota G, Cesaro P, Martino A, Zuccala G, Cianci R, Nista E, Larocca LM, Vecchio FM, Gasbarrini A, Gasbarrini G. High accuracy and cost-effectiveness of a biopsy-avoiding endoscopic approach in diagnosing coeliac disease. Aliment Pharmacol Ther. 2006 Jan 1;23(1):61-9. doi: 10.1111/j.1365-2036.2006.02732.x. PMID 16393281
- [Background] Vogelsang H, Hanel S, Steiner B, Oberhuber G. Diagnostic duodenal bulb biopsy in celiac disease. Endoscopy. 2001 Apr;33(4):336-40. doi: 10.1055/s-2001-13702. PMID 11315895
- [Background] Cammarota G, Pirozzi GA, Martino A, Zuccala G, Cianci R, Cuoco L, Ojetti V, Landriscina M, Montalto M, Vecchio FM, Gasbarrini G, Gasbarrini A. Reliability of the "immersion technique" during routine upper endoscopy for detection of abnormalities of duodenal villi in patients with dyspepsia. Gastrointest Endosc. 2004 Aug;60(2):223-8. doi: 10.1016/s0016-5107(04)01553-6. PMID 15278049
- [Background] Cammarota G, Cesaro P, La Mura R, Martino A, Cazzato A, Miele L, Lupascu A, Vecchio FM, Larocca LM, Grieco A, Gasbarrini G. Role of the "immersion technique" in diagnosing celiac disease with villous atrophy limited to the duodenal bulb. J Clin Gastroenterol. 2007 Jul;41(6):571-5. doi: 10.1097/01.mcg.0000225625.99415.c0. PMID 17577113
- [Background] Badreldin R, Barrett P, Wooff DA, Mansfield J, Yiannakou Y. How good is zoom endoscopy for assessment of villous atrophy in coeliac disease? Endoscopy. 2005 Oct;37(10):994-8. doi: 10.1055/s-2005-870245. PMID 16189773
- [Background] Niveloni S, Fiorini A, Dezi R, Pedreira S, Smecuol E, Vazquez H, Cabanne A, Boerr LA, Valero J, Kogan Z, Maurino E, Bai JC. Usefulness of videoduodenoscopy and vital dye staining as indicators of mucosal atrophy of celiac disease: assessment of interobserver agreement. Gastrointest Endosc. 1998 Mar;47(3):223-9. doi: 10.1016/s0016-5107(98)70317-7. PMID 9580349
- [Background] Kiesslich R, Mergener K, Naumann C, Hahn M, Jung M, Koehler HH, Nafe B, Kanzler S, Galle PR. Value of chromoendoscopy and magnification endoscopy in the evaluation of duodenal abnormalities: a prospective, randomized comparison. Endoscopy. 2003 Jul;35(7):559-63. doi: 10.1055/s-2003-40240. PMID 12822089
- [Background] Siegel LM, Stevens PD, Lightdale CJ, Green PH, Goodman S, Garcia-Carrasquillo RJ, Rotterdam H. Combined magnification endoscopy with chromoendoscopy in the evaluation of patients with suspected malabsorption. Gastrointest Endosc. 1997 Sep;46(3):226-30. doi: 10.1016/s0016-5107(97)70091-9. PMID 9378209
- [Background] Lo A, Guelrud M, Essenfeld H, Bonis P. Classification of villous atrophy with enhanced magnification endoscopy in patients with celiac disease and tropical sprue. Gastrointest Endosc. 2007 Aug;66(2):377-82. doi: 10.1016/j.gie.2007.02.041. PMID 17643717
- [Background] Cammarota G, Cesaro P, Cazzato A, Fedeli P, Sparano L, Vecchio FM, Larocca LM, Gasbarrini G. Optimal band imaging system: a new tool for enhancing the duodenal villous pattern in celiac disease. Gastrointest Endosc. 2008 Aug;68(2):352-7. doi: 10.1016/j.gie.2008.02.054. Epub 2008 Jun 11. PMID 18547574
- [Background] Cammarota G, Ianiro G, Sparano L, La Mura R, Ricci R, Larocca LM, Landolfi R, Gasbarrini A. Image-enhanced endoscopy with I-scan technology for the evaluation of duodenal villous patterns. Dig Dis Sci. 2013 May;58(5):1287-92. doi: 10.1007/s10620-012-2467-y. Epub 2012 Oct 31. PMID 23108566
- [Background] Gheorghe C. Narrow-band imaging endoscopy for diagnosis of malignant and premalignant gastrointestinal lesions. J Gastrointestin Liver Dis. 2006 Mar;15(1):77-82. PMID 16680239
- [Background] Banerjee R, Reddy DN. High-resolution narrow-band imaging can identify patchy atrophy in celiac disease: targeted biopsy can increase diagnostic yield. Gastrointest Endosc. 2009 Apr;69(4):984-5. doi: 10.1016/j.gie.2008.07.012. No abstract available. PMID 19327498
- [Background] Singh R, Nind G, Tucker G, Nguyen N, Holloway R, Bate J, Shetti M, George B, Tam W. Narrow-band imaging in the evaluation of villous morphology: a feasibility study assessing a simplified classification and observer agreement. Endoscopy. 2010 Nov;42(11):889-94. doi: 10.1055/s-0030-1255708. Epub 2010 Nov 11. PMID 21072704
- [Background] De Luca L, Ricciardiello L, Rocchi MB, Fabi MT, Bianchi ML, de Leone A, Fiori S, Baroncini D. Narrow band imaging with magnification endoscopy for celiac disease: results from a prospective, single-center study. Diagn Ther Endosc. 2013;2013:580526. doi: 10.1155/2013/580526. Epub 2013 Aug 6. PMID 23983448
- [Background] Goswami A, Dadhich S, Bhargava N. Use of narrow band imaging in assessing duodenal villous atrophy. Indian J Gastroenterol. 2014 Sep;33(5):440-4. doi: 10.1007/s12664-014-0489-4. Epub 2014 Jul 13. PMID 25015746
- [Background] Oxentenko AS, Grisolano SW, Murray JA, Burgart LJ, Dierkhising RA, Alexander JA. The insensitivity of endoscopic markers in celiac disease. Am J Gastroenterol. 2002 Apr;97(4):933-8. doi: 10.1111/j.1572-0241.2002.05612.x. PMID 12003429
- [Derived] Gulati S, Emmanuel A, Ong M, Pavlidis P, Patel M, El-Menabawey T, Vackova Z, Dubois P, Murino A, Martinek J, Sethi A, Neumann H, Haji A, Hayee B. Near-focus narrow-band imaging classification of villous atrophy in suspected celiac disease: development and international validation. Gastrointest Endosc. 2021 Dec;94(6):1071-1081. doi: 10.1016/j.gie.2021.06.031. Epub 2021 Jul 3. PMID 34228981